CLINICAL TRIAL: NCT01032889
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study of ATX-101 (Sodium Deoxycholate Injection) Versus Placebo for the Reduction of Localized Subcutaneous Fat in the Submental Area (SMF) Using Magnetic Resonance Imaging (MRI) and a Battery of Clinician- and Subject-reported Measurements.
Brief Title: Deoxycholic Acid Injection Submental Fat (SMF) Magnetic Resonance Imaging (MRI) and Subject-reported Outcome Measures Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-101-09-15
Record Dates: First submitted 2009-12-10; First posted 2009-12-16 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Moderate or Severe Submental Fullness
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Deoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo administered in 0.2 mL injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Placebo
- Deoxycholic acid Injection 1 mg/cm² (Experimental): Participants received deoxycholic acid 1 mg/cm² administered in 0.2 mL injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Deoxycholic acid injection
- Deoxycholic acid Injection 2 mg/cm² (Experimental): Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Deoxycholic acid injection

INTERVENTIONS:
Drug: Deoxycholic acid injection
  Other Names: ATX-101; Kybella
  Arms: Deoxycholic acid Injection 1 mg/cm²; Deoxycholic acid Injection 2 mg/cm²
Drug: Placebo — Phosphate buffered saline placebo for injection
  Arms: Placebo

SUMMARY:
Evaluation of the safety, tolerability and efficacy of deoxycholic acid injection in the reduction of submental fat (fat below the chin).

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe submental fat
* Dissatisfaction with submental area
* History of stable body weight
* Signed informed consent

Exclusion Criteria:

* Any medical or other condition that would affect subject safety or evaluation of efficacy
* Previous intervention in the submental area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, MD, PhD, Study Director — Kythera Biopharmaceuticals, Inc.
Locations (9):
- United States (9):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Beverly Hills, California
  - Investigational Site, San Francisco, California
  - Investigational Site, Naperville, Illinois
  - Investigational Site, Chestnut Hill, Massachusetts
  - Investigational Site, Fridley, Minnesota
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Omaha, Nebraska
  - Investigational Site, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 centers in the United States.
Period: Overall Study
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Started | 41 | 43 | 45
Received Treatment | 41 | 43 | 45
Completed | 33 | 28 | 42
Not Completed | 8 | 15 | 3
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Withdrawal of Consent | 1 | 2 | 1
Not completed — Patient Request | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Lack of Submental Fat | 2 | 8 | 1
Not completed — Miscellaneous Reasons | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo | Total
Number analyzed (Participants) | 41 | 43 | 45 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (9.57) | 45.6 (9.43) | 47.4 (10.20) | 46.1 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 31 | 92
  Male | 12 | 11 | 14 | 37
Race/Ethnicity, Customized [Number; unit: participants] — Participants could select more than one category.
  participants
    White | 38 | 35 | 36 | 109
    Hispanic or Latino | 1 | 6 | 4 | 11
    Black or African American | 3 | 2 | 2 | 7
    Asian | 1 | 0 | 2 | 3
    Other | 1 | 1 | 1 | 3
Weight [Mean (Standard Deviation); unit: kg] — Data available for 40, 43 and 45 participants in each treatment arm respectively.
  kg | 84.88 (15.835) | 89.32 (21.225) | 87.78 (16.059) | 87.39 (17.851)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Data available for 40, 43 and 45 participants in each treatment arm respectively.
  kg/m² | 29.68 (4.845) | 31.48 (6.633) | 30.85 (5.315) | 30.70 (5.665)
Fitzpatrick Skin Type [Number; unit: participants] — Fitzpatrick Skin Type is a numerical classification schema for human skin color and typical response to ultraviolet (UV) light:
  * Type I: Pale white skin, blue/hazel eyes, blond/red hair; Always burns, does not tan.
  * Type II: Fair skin, blue eyes; Burns easily, tans poorly.
  * Type III: Darker white skin; Tans after initial burn.
  * Type IV: Light brown skin; Burns minimally, tans easily.
  * Type V: Brown skin; Rarely burns, tans darkly easily.
  * Type VI: Dark brown or black skin; Never burns, always tans darkly.
  participants
    I - III | 30 | 26 | 33 | 89
    IV - VI | 11 | 17 | 12 | 40
Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) Rating [Number; unit: participants] — CR-SMFRS Ratings:
  * 0 = Absent submental convexity: No localized submental fat evident;
  * 1 = Mild submental convexity: Minimal, localized submental fat;
  * 2 = Moderate submental convexity: Prominent, localized submental fat;
  * 3 = Severe submental convexity: Marked, localized submental fat;
  * 4 = Extreme submental convexity.
  participants
    2 | 17 | 22 | 18 | 57
    3 | 24 | 21 | 27 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician-Reported Submental Fat Rating Scale Scores
Description: The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0-4) with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 weeks after last treatment (up to 32 weeks after first treatment)
Population: Modified Intent-to-Treat (mITT) population including all randomized participants who received at least 1 injection of study drug and had at least 1 post-baseline observation for CR-SMFRS, Subject Self-Rating Scale (SSRS), or magnetic resonance imaging (MRI) volume. Last observation carried forward (LOCF) method was used to impute missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 40 | 42 | 45
units on a scale | -0.7 [-0.90 to -0.45] | -0.8 [-1.06 to -0.62] | -0.4 [-0.58 to -0.16]
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; There was no formal hypothesis testing and no adjustments for multiple comparisons; Test type: Superiority or Other; p = 0.052, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -0.3, 95% CI 2-sided [-0.61 to 0.00]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; There was no formal hypothesis testing and no adjustments for multiple comparisons; Test type: Superiority or Other; p = 0.003, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -0.5, 95% CI 2-sided [-0.77 to -0.16]

2. Primary Outcome: Change From Baseline in Patient-Reported Submental Fat Scale Rating Scale (PR-SMFRS)
Description: The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" answered on a 5-point ordinal scale (0-4) with 0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 weeks after last treatment (up to 32 weeks after first treatment)
Population: Modified intent-to-treat population with available Baseline data; LOCF method was used to impute missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 37 | 39 | 43
units on a scale | -0.9 [-1.17 to -0.72] | -1.3 [-1.53 to -1.09] | -0.7 [-0.91 to -0.49]
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; There was no formal hypothesis testing and no adjustments for multiple comparisons; Test type: Superiority or Other; p = 0.117, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -0.2, 95% CI 2-sided [-0.55 to 0.06]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; There was no formal hypothesis testing and no adjustments for multiple comparisons; Test type: Superiority or Other; p < 0.001, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -0.6, 95% CI 2-sided [-0.91 to -0.30]

3. Primary Outcome: Change From Baseline in Patient-Reported Submental Fat Impact Scale (PR-SMFIS)
Description: The PR-SMFIS assesses the impact of submental fat on self-perception of 6 emotional and visual characteristics related to the appearance of submental fullness (unhappy, bothered, self-conscious, embarrassed, look older, and look overweight) as evaluated by the participant. Each item is rated on an 11-point numeric scale from 0 to 10. Scores for the 6 items were averaged to generate a PR-SMFIS total scale score ranging from 0 to 10 where 0 is a positive outcome and 10 is a negative outcome. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 weeks after last treatment (up to 32 weeks after first treatment)
Population: Modified intent-to-treat population with available Baseline data; LOCF method was used to impute missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 39 | 40 | 44
units on a scale | -3.5 [-4.21 to -2.78] | -4.5 [-5.25 to -3.81] | -2.1 [-2.73 to -1.37]
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; There was no formal hypothesis testing and no adjustments for multiple comparisons; Test type: Superiority or Other; p = 0.005, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -1.4, 95% CI 2-sided [-2.44 to -0.46]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; There was no formal hypothesis testing and no adjustments for multiple comparisons; Test type: Superiority or Other; p < 0.001, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -2.5, 95% CI 2-sided [-3.48 to -1.48]

4. Secondary Outcome: Change From Baseline in Submental Fat Volume
Description: Submental fat volume was measured by magnetic resonance imaging (MRI).
Time Frame: Baseline and 12 weeks after last treatment (up to 32 weeks after first treatment)
Population: Modified intent-to-treat population; LOCF method was used to impute missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm³
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 40 | 42 | 45
mm³ | -614 [-1093 to -136] | -118 [-644 to 407] | -8.1 [-742 to 725.7]
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.166, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -606, 95% CI 2-sided [-1482 to 269.3]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.803, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -110, 95% CI 2-sided [-1013 to 792.6]

5. Secondary Outcome: Change From Baseline in Submental Fat Thickness
Description: Submental fat thickness was measured by magnetic resonance imaging (MRI).
Time Frame: Baseline and 12 weeks after last treatment (up to 32 weeks after first treatment)
Population: Modified intent-to-treat population; LOCF method was used to impute missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 40 | 42 | 45
mm | -1.8 [-2.37 to -1.19] | -1.9 [-2.51 to -1.35] | -0.3 [-0.83 to 0.29]
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -1.5, 95% CI 2-sided [-2.32 to -0.69]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; The ANCOVA model included terms for treatment group and the baseline covariate; Difference from placebo = -1.7, 95% CI 2-sided [-2.46 to -0.85]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 12 weeks after the last dose (up to 32 weeks after first treatment).
Description: The safety population included all participants who received at least one injection of study drug.
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/43 | 0/45
Other Adverse Events (participants affected / at risk) | 40/41 | 40/43 | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid Injection 1 mg/cm² (N=41) | Deoxycholic Acid Injection 2 mg/cm² (N=43) | Placebo (N=45)
Intracranial hypotension (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid Injection 1 mg/cm² (N=41) | Deoxycholic Acid Injection 2 mg/cm² (N=43) | Placebo (N=45)
Injection site anesthesia (General disorders) | 26 | 26 | 4
Injection site discomfort (General disorders) | 3 | 2 | 0
Injection site edema (General disorders) | 19 | 16 | 13
Injection site erythema (General disorders) | 15 | 12 | 14
Injection site hematoma (General disorders) | 23 | 21 | 31
Injection site hemorrhage (General disorders) | 3 | 1 | 7
Injection site induration (General disorders) | 11 | 14 | 5
Injection site nodule (General disorders) | 5 | 4 | 2
Injection site pain (General disorders) | 29 | 23 | 13
Injection site paresthesia (General disorders) | 7 | 4 | 3
Injection site pruritus (General disorders) | 11 | 11 | 3
Injection site swelling (General disorders) | 16 | 17 | 5
Nasopharyngitis (Infections and infestations) | 6 | 4 | 7
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 3 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Study Agreement requires that the investigator or institution obtain written consent from Kythera prior to presenting and/or publishing results of this study.